CLINICAL TRIAL: NCT05575206
Title: Untersuchung Des Einflusses Von Genetischen Varianten in ELAPOR1 Oder ELAPOR2 Auf Die Insulinsekretion Und Glukoseregulation im Menschen
Brief Title: The Influence of Genetic Variations in ELAPOR1 or ELAPOR2 on Insulin Secretion and Glucose Regulation in Humans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: INCEPTOR
Record Dates: First submitted 2022-09-26; First posted 2022-10-12 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes; Impaired Insulin Secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genetic analysis of ELAPOR1 and ELAPOR2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rare genetic variant in ELAPOR1 or ELAPOR2: Patients undergo several examinations. Beside anthropometric measurements, bioelectrical impedance analysis, an 2h-oral glucose tolerance test (OGTT) and a hyperglycemic clamp is performed.

SUMMARY:
Insulin resistance and the depletion of insulin secretion are major pathogenetic aspects of type 2 diabetes mellitus. Recently, inceptor, a receptor on the surface of beta cells was dicovered. Inceptor promotes beta cell resistance to insulin and IGF-1.

In humans, the inceptor is encoded by the two genes ELAPOR1 and ELAPOR2. Whether functional mutations in these genes affect insulin secretion and glucose regulation in humans has not been investigated so far.

In this study we investigate the influence of genetic variations in ELAPOR1 or ELAPOR2 on insulin secretion and glucose regulation in humans by hygerglycemic glucose clamp technique and oral glucose tolerance test respectively.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a heterogenic disorder with a complex pathogenesis. Although, loss of beta cell function is crucial for the manifestation of the disease. Genome-wide association studies identified more than 400 genetic variations associated with a reduced beta cell function. Interestingly, beta cells are not only responsible for the secretion of insulin, but are also insulin sensitive cells, whereby insulin secretion and proliferation is regulated. It is well known that an insulin and insulin-like growth factor (IGF-1) resistance lead to the manifestation of type 2 diabetes. Underlying mechanism are mostly unknown. Recently, a new receptor on the surface of beta-cells was identified which mediates the resistance of beta cells to insulin and IGF-1. This insulin inhibitory receptor (Inceptor) induces its inhibitory function via clathrin-mediated endocytosis of the INSR-IGF-1R complex. In mice, inceptor is encoded by lir and its knock-out leads to beta cell proliferation and an increased insulin secretion. In animal models, treatment with monoclonal antibodies against the extracellular domain of inceptor, leads to a significantly improved glucose regulation. Thus, pharmacological interventions on the inceptor could represent a novel therapeutic approach for the treatment of type 2 diabetes mellitus. In humans, inceptor is encoded by genes ELAPOR1 and ELAPOR2. So far, there are no studies in humans that investigate if functional mutations in these genes affect insulin secretion and glucose regulation. The aim of this study is to investigate, whether subjects with genetic variants in ELAPOR1 or ELAPOR2 have altered insulin secretion and thus altered glucose regulation. For this purpose, the study results are compared with a reference cohort without variants in ELAPOR1 or ELAPOR2 (matched for age, sex, waist to hip ratio and BMI) from our databases of previous studies (e.g. PLIS: NCT01947595, PREG: NCT04270578, KNOMA: NCT04950283). Insulin secretion is assessed by hyperglycemic glucose clamp technique. An oral glucose tolerance test will be performed to assess glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* subjects with genetic variations in ELAPOR1 and ELAPOR2

Exclusion Criteria:

* Women during pregnancy and lactation
* Treatment with any medication effecting on glucose metabolism like anti-diabetic drugs or steroids
* Any pancreatic disease
* Known current presence or history of severe neurological or psychiatric diseases, schizophrenia, bipolar disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with genetic variations in ELAPOR1 and ELAPOR2
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion capacity | -15 minutes - 130 minutes
  Glucose stimulated insulin secretion adjusted for insulin sensitivity during an hyperglycemic clamp in subjects with genetic variants in ELAPOR1 and ELAPOR2 compared to a control cohort without genetic variants.

SECONDARY OUTCOMES:
Glucose tolerance status | 0-120 minutes
  Glucose tolerance status examined by 2h-oral glucose tolerance test in subjects with genetic variants in ELAPOR1 and ELAPOR2 compared to a control cohort without genetic variants.

CONTACTS AND LOCATIONS:
Overall Officials: Reiner Jumpertz-von Schwartzenberg, MD, Principal Investigator — University Hopsital Tübingen
Locations (1):
- University Hopsital Tübingen, Tübingen, Germany